CLINICAL TRIAL: NCT05003674
Title: A Feasibility, Prospective, Multi-centre, Repeated-measures Study Evaluating the Performance of Focused Multipolar Stimulation in Adult Cochlear Implant Recipients
Brief Title: A Feasibility Study Evaluating the Performance of Focused Multipolar Stimulation in Adult Cochlear Implant Recipients
Acronym: FOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AI5782
Record Dates: First submitted 2021-07-21; First posted 2021-08-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Hearing Impairment
Keywords: cochlear implantation
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adults cochlear implant recipients receiving alternative stimulation strategy (Experimental): ACE strategy, 8 maxima, alternative mode
  Interventions: Device: Focused stimulation strategy
- Adults cochlear implant recipients receiving Standard-of-Care stimulation strategy. (Active Comparator): ACE strategy, 8 maxima, monopolar mode.
  Interventions: Device: ACE stimulation strategy

INTERVENTIONS:
Device: Focused stimulation strategy — Investigational focused stimulation strategy
  Arms: Adults cochlear implant recipients receiving alternative stimulation strategy
Device: ACE stimulation strategy — Standard of care stimulation strategy
  Arms: Adults cochlear implant recipients receiving Standard-of-Care stimulation strategy.

SUMMARY:
This feasibility study is designed to explore several facets of hearing performance that may show improvements for alternative modes of stimulation compared to Monopolar (MP) stimulation within a group of adult cochlear-implant recipients. Measures of speech recognition, music appreciation, listening effort, quality of life, and real-world assessments will be gathered to determine the most promising benefits for further examination.

DETAILED DESCRIPTION:
Alternative modes of stimulation will be investigated that may improve spectral resolution through reduced cochlear spread of excitation and in turn provide enhanced speech perception and real-world clinical benefits over MP stimulation. The purpose of this feasibility study is to explore several facets of hearing performance that may show improvements with these alternative modes of stimulation compared to MP stimulation within a group of adult cochlear-implant recipients. Measures of speech recognition, music appreciation, listening effort, quality of life, and real-world assessments will be gathered to determine the most promising benefits for further examination. Individual neural, psychophysical, cognitive, and electrode placement data will also be obtained to inform questions related to across-subject variability, and practical aspects of power consumption and device fitting will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older.
2. Candidate for unilateral cochlear implant with Slim Modiolar electrode array as determined by the implanting centre.
3. English spoken as a primary language.
4. Willingness to comply with all investigational requirements.
5. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Previous or existing cochlear-implant recipient.
2. Evidence of severe or greater sensorineural hearing loss prior to five years of age.
3. Open-set pre-operative word score > 70% in the contralateral ear.
4. Duration of severe to profound hearing loss > 20 years in the ear to be implanted.
5. Adults with functional acoustic hearing in the ear to be implanted who desire to use an acoustic component in the implanted ear.
6. Ossification or other cochlear anomaly that might prevent complete insertion of the electrode array.
7. Hearing loss of neural or central origin.
8. Medical or psychological conditions that would contraindicate undergoing surgery.
9. Women who are pregnant.
10. Additional handicaps that would prevent or restrict participation in the audiological evaluations.
11. Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and prosthetic device.
12. Inability or unwillingness to use a hand-held device to control the sound processor and to collect test and survey data.
13. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
14. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
15. Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
16. Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Mean difference between stimulation modes for sentence perception in background noise (dB) (AuSTIN) | 7 months

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - NextSense - Deakin, Deakin, Australian Capital Territory
  - NextSense - Broadmeadow, Broadmeadow, New South Wales
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
  - St Vincent's Private Hospital, East Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No